CLINICAL TRIAL: NCT01638559
Title: Immunosuppression Withdrawal for Stable Pediatric Liver Transplant Recipients
Acronym: iWITH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT iWITH; U01AI100807 (NIH); RTB-001 (Other: DAIT NIAID); NIAID DAIT CRMS ID#: 20129 (Other: DAIT NIAID)
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-09

CONDITIONS: Liver Transplant Recipients; Liver Transplantation; Immunosuppression
Keywords: liver transplant; allograft function; anti-rejection; immunosuppression withdrawal; tolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Immunosuppression withdrawal (Experimental): Gradual withdrawal of immunosuppressive treatment withdrawal as per protocol.
  Interventions: Drug: Immunosuppression withdrawal

INTERVENTIONS:
Drug: Immunosuppression withdrawal — Participants will undergo gradual ISW in no less than 36 weeks and no more than 52 weeks with frequent monitoring of liver tests. All participants will be followed for 48 months ensuring a minimum of 36 months of follow-up after successful ISW.
  Other Names: ISW

SUMMARY:
The primary objective of this study is to assess the efficacy of immunosuppression withdrawal (ISW) in pediatric liver transplant (tx) recipients.

DETAILED DESCRIPTION:
Anti-rejection medicines, also known as immunosuppressive drugs, are prescribed to organ transplant recipients to prevent rejection of the new organ. Long-term use of these medicines places transplant recipients at higher risk of serious infections and certain types of cancer.

This study seeks to:

* Find out if it is safe to slowly reduce and then completely stop the immunosuppression taken by children who have received liver transplants. This process is called 'immunosuppression withdrawal'or ISW.
* Find blood or liver biopsy tests that can help transplant doctors in the future to predict if it is safe to decrease or stop immunosuppression drugs in children who have had a liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or parent guardian must be able to understand and provide informed consent;
* Is the recipient of a living or deceased donor liver tx when subject was less than or equal to 6 years of age;
* Is at least 4 years post-tx at the time of study enrollment;
* Has normal allograft function defined as Alanine aminotransferase (ALT) < 50 IU/l and gamma-glutamyl transferase (GGT) < 50 IU/l;
* Has no evidence of acute rejection (AR) or chronic rejection (CR) within the past 2 years, based on medical history;
* Is stable on IS monotherapy with a calcineurin inhibitor (CNI);
* For female subjects of childbearing potential, subject must have a negative pregnancy test upon study entry;
* For female and male subjects with reproductive potential, subject must agree to use FDA approved methods of birth control for the duration of the study;
* Must be negative for hepatitis B virus (HBV) and hepatitis C virus (HCV) infection within one year of enrollment;
* Must have screening biopsy that fulfills, based on central pathology reading, the following criteria:

  * Portal inflammation and interface activity: Preferably absent, but minimal to focal mild portal mononuclear inflammation may be present. Interface necro-inflammatory activity is absent or equivocal/minimal and, if present, involves a minority of portal tracts.
  * Centrizonal/peri-venular inflammation: Preferably absent, but minimal to focal mild perivenular mononuclear inflammation may be present. Perivenular necro-inflammatory activity is absent or equivocal/minimal and, if present, involves a minority of terminal hepatic venules.
  * Bile duct changes: No lymphocytic bile duct damage, ductopenia and biliary epithelial senescence changes, unless there is an alternative, non-immunologic explanation (e.g. biliary strictures).
  * Fibrosis: < Ishak Stage 3 (i.e. not more than occasional portal-to-portal bridging). Perivenular fibrosis should be less than "moderate", according to Banff Criteria.
  * Arteries: Negative for obliterative or foam cell arteriopathy.

Exclusion Criteria:

* Have received a liver tx for autoimmune liver disease, including autoimmune hepatitis or primary sclerosing cholangitis;
* Have received a liver tx for hepatitis B or hepatitis C;
* Have received a second organ transplant before, simultaneously, or after liver tx;
* Have a calculated glomerular filtration rate (modified Schwartz formula) of less than 60 mL/min/1.73 m^2;
* Have had a 50 percent (%) dose increase in CNI within 6 months of screening;
* Have discontinued a second IS agent within 12 months of screening;
* Have any systemic illness requiring or likely to require chronic or recurrent use of IS;
* Is pregnant or breastfeeding;
* Is unwilling or unable to adhere with study requirements and procedures;
* Have mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements;
* Is unwilling or unable to provide consent or comply with the study protocol;
* Has used investigational drugs within 4 weeks of enrollment;
* Is receiving treatment for HIV infection;
* Has received any licensed or investigational live attenuated vaccine(s) within two months of enrollment;
* Has any medical condition that, in the opinion of the investigator, will interfere with safe participation in the trial.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 161 (Actual)
Dates: Start 2012-08-14 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2018-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S Feng, M.D., Ph.D., Principal Investigator — University of California, San Francisco; J Bucuvalas, M.D., Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (12):
- United States (11):
  - University of California, San Francisco, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Emory University and Children's Hospital of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Michigan C. S. Mott Children's Hospital, Ann Arbor, Michigan
  - St. Louis Children's Hospital - Washington University, St Louis, Missouri
  - New York Presbyterian Morgan Stanley Children's Hospital - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in ImmPort, a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: The aim is to share data available to the public within 24 months upon completion of the study.
Access Criteria: ImmPort public data access.
URL: https://immport.niaid.nih.gov/

REFERENCES:
- [Background] Feng S, Ekong UD, Lobritto SJ, Demetris AJ, Roberts JP, Rosenthal P, Alonso EM, Philogene MC, Ikle D, Poole KM, Bridges ND, Turka LA, Tchao NK. Complete immunosuppression withdrawal and subsequent allograft function among pediatric recipients of parental living donor liver transplants. JAMA. 2012 Jan 18;307(3):283-93. doi: 10.1001/jama.2011.2014. PMID 22253395
- [Background] Perito ER, Mohammad S, Rosenthal P, Alonso EM, Ekong UD, Lobritto SJ, Feng S. Posttransplant metabolic syndrome in the withdrawal of immunosuppression in Pediatric Liver Transplant Recipients (WISP-R) pilot trial. Am J Transplant. 2015 Mar;15(3):779-85. doi: 10.1111/ajt.13024. Epub 2015 Feb 3. PMID 25648649
- [Background] Reding R. Long-term complications of immunosuppression in pediatric liver recipients. Acta Gastroenterol Belg. 2005 Oct-Dec;68(4):453-6. PMID 16433002
- [Derived] Wood-Trageser MA, Lesniak D, Gambella A, Golnoski K, Feng S, Bucuvalas J, Sanchez-Fueyo A, Demetris AJ. Next-generation pathology detection of T cell-antigen-presenting cell immune synapses in human liver allografts. Hepatology. 2023 Feb 1;77(2):355-366. doi: 10.1002/hep.32666. Epub 2022 Aug 1. PMID 35819312
- [Derived] Mohammad S, Sundaram SS, Mason K, Lobritto S, Martinez M, Turmelle YP, Bucuvalas J, Feng S, Alonso EM. Improvements in Disease-Specific Health-Related Quality of Life of Pediatric Liver Transplant Recipients During Immunosuppression Withdrawal. Liver Transpl. 2021 May;27(5):735-746. doi: 10.1002/lt.25963. PMID 33280227
- [Derived] Feng S, Bucuvalas JC, Mazariegos GV, Magee JC, Sanchez-Fueyo A, Spain KM, Lesniak A, Kanaparthi S, Perito E, Venkat VL, Burrell BE, Alonso EM, Bridges ND, Doo E, Gupta NA, Himes RW, Ikle D, Jackson AM, Lobritto SJ, Jose Lozano J, Martinez M, Ng VL, Rand EB, Sherker AH, Sundaram SS, Turmelle YP, Wood-Trageser M, Demetris AJ. Efficacy and Safety of Immunosuppression Withdrawal in Pediatric Liver Transplant Recipients: Moving Toward Personalized Management. Hepatology. 2021 May;73(5):1985-2004. doi: 10.1002/hep.31520. PMID 32786149
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Immune Tolerance Network (ITN) — http://www.immunetolerance.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 161 participants were enrolled (11 sites in the US,1 site in Canada) between August 2012 and April 2014. N=88 of the enrolled participants were eligible to initiate immunosuppression withdrawal (ISW) and the remaining N=73 participants were terminated (e.g., ineligible to proceed with ISW) based on biopsy findings or other pre-specified criteria.
Pre-assignment Details: Informed consent was obtained from eligible individuals who then underwent a study-mandated biopsy to determine if they were eligible to initiate immunosuppression withdrawal, based on pre-specified histologic and other criteria.
Groups:
- Participants That Initiated Immunosuppression Withdrawal (ISW): Pediatric liver transplant recipients with stable liver tests (ALT and GGT), no evidence of rejection in the preceding 2 years, and at least 4 years post-transplant, and a qualifying liver biopsy at screening underwent gradual Immunosuppression withdrawal in no less than 36 weeks and no more than 52 weeks with frequent monitoring of liver tests. All participants were followed for 48 months ensuring a minimum of 36 months of follow-up after successful Immunosuppression withdrawal..
Period: Overall Study
Arm/Group | Participants That Initiated Immunosuppression Withdrawal (ISW)
Started | 88
Completed | 85 (Completion through the time of the primary endpoint (outcome).)
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Not completed — Subject declined to travel for biopsy | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat
Arm/Group | Participants That Initiated Immunosuppression Withdrawal (ISW)
Number analyzed (Participants) | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 88
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 74
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 76
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  Canada | 6
  United States | 82
Entry Calcineurin Inhibitor (CNI) Daily Dose [Mean (Standard Deviation); unit: mg] — Dose of either Cyclosporine or Tacrolimus that the participant was on prior to Initiation of Immunosuppression Withdrawal (ISW). Population: 7 participants were on Cyclosporine, and 81 were on Tacrolimus for Immunosuppression, for a total of 88 analyzed participants.
  mg
    Cyclosporine: number analyzed (Participants) | 7
    Cyclosporine | 65.7 (22.99)
    Tacrolimus: number analyzed (Participants) | 81
    Tacrolimus | 2.1 (1.33)
Screening Biopsy Ishak Stage [Count of Participants; unit: Participants] — Ishak Stage from Screening Liver Biopsy (higher score indicates more severe liver fibrosis) 0=No fibrosis; 1=Fibrous expansion of some portal areas, with or without short fibrous septa; 2=Fibrous expansion of most portal areas, with or without short fibrous septa; 3=Fibrous expansion of most portal areas with occasional portal to portal bridging; 4=Fibrous expansion of portal areas with marked bridging (portal to portal) as well as portal to central; 5=Marked bridging (portal to portal and/or portal to central) with occasional nodules (incomplete cirrhosis); 6=Cirrhosis, probable or definite
  Participants
    0 | 19
    1 | 57
    2 | 12
Screening Child Health Related Quality of Life Scores on a Scale [Mean (Standard Deviation); unit: Quality of Life Scores on a Scale] — Health related quality of life was measured by the PedsQL 4.0 Generic Core scale, the Multidimensional Fatigue scale, and the PedsQL 3.0 Transplant module. Each score ranges from 0-100, with a higher score indicating a better quality of life. Measure is broken down by Operationally Tolerant Participants (Tolerant), Operationally Non-Tolerant Participants (Non-Tolerant), and Total Participants (All Participants). Population: Number of Participants Analyzed added for each row.
  Quality of Life Scores on a Scale
    All Participants - Total Generic Score | 80.7 (13.69)
    All Participants - Total Fatigue Score | 74.9 (17.75)
    All Participants - Total Transplant Score | 85.6 (9.54)
    Tolerant Participants - Total Generic Score: number analyzed (Participants) | 33
    Tolerant Participants - Total Generic Score | 80.7 (14.59)
    Tolerant Participants - Total Fatigue Score: number analyzed (Participants) | 33
    Tolerant Participants - Total Fatigue Score | 75.6 (15.82)
    Tolerant Participants - Total Transplant Score: number analyzed (Participants) | 33
    Tolerant Participants - Total Transplant Score | 86.0 (10.16)
    Non-Tolerant Participants - Total Generic Score: number analyzed (Participants) | 55
    Non-Tolerant Participants - Total Generic Score | 80.6 (13.26)
    Non-Tolerant Participants - Total Fatigue Score: number analyzed (Participants) | 55
    Non-Tolerant Participants - Total Fatigue Score | 74.5 (18.94)
    Non-Tolerant Participants - Total Transplant Score: number analyzed (Participants) | 55
    Non-Tolerant Participants - Total Transplant Score | 85.4 (9.27)

OUTCOME MEASURES:

1. Primary Outcome: Number of Operationally Tolerant Participants
Description: Number of participants that are operationally tolerant, defined as those who successfully withdraw from immunosuppression and maintain normal allograft status as assessed by liver biopsy and liver tests 12 months after complete immunosuppression withdrawal.
Time Frame: 12 Months after complete immunosuppression withdrawal
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Participants That Initiated Immunosuppression Withdrawal (ISW)
Number analyzed (Participants) | 88
Participants | 33

2. Secondary Outcome: Number of Participants With Clinical Complications Usually Attributed to Immunosuppression
Description: This composite endpoint is comprised of clinical complications related to immunosuppression withdrawal and is defined as the occurrence of any of the following: death or graft loss, histologic evidence of refractory acute rejection or biopsy confirmed chronic rejection (CR).
Time Frame: Time from immunosuppression withdrawal through a minimum of 36 months and a maximum of 48 months of follow-up
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Participants That Initiated Immunosuppression Withdrawal (ISW)
Number analyzed (Participants) | 88
Participants | 0

3. Secondary Outcome: Time to Increased Immunosuppression or Re-Initiation of Immunosuppression
Description: The median time (in days) from start of withdrawal from immunosuppression drugs to increasing or re-starting immunosuppression.
Time Frame: Time from immunosuppression withdrawal through a minimum of 36 months and maximum of 48 months of follow-up
Population: Participants that either restarted immunosuppression or increased their dose of immunosuppression
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Participants That Increased IS Dosing or Restarted IS: Pediatric liver transplant recipients with stable liver tests (ALT and GGT), no evidence of rejection in the preceding 2 years, and at least 4 years post-transplant, and a qualifying liver biopsy at screening underwent gradual Immunosuppression (IS) withdrawal in no less than 36 weeks and no more than 52 weeks with frequent monitoring of liver tests. All participants were followed for 48 months ensuring a minimum of 36 months of follow-up after successful IS withdrawal. These participants either failed IS withdrawal or restarted IS after completing withdrawal.
Arm/Group | Participants That Increased IS Dosing or Restarted IS
Number analyzed (Participants) | 50
days | 204 [167 to 246]

4. Secondary Outcome: Time to Resolution of Rejection
Description: The median time (in weeks) from biopsy proven rejection to resolution of rejection defined as both liver function tests Alanine Aminotransferase (ALT) and Gamma-Glutamyl Transferase (GGT) returning to ≤ 1.5 the baseline values.
Time Frame: Time from immunosuppression withdrawal through a minimum of 36 months and maximum of 48 months of follow-up
Population: Intent-to-Treat
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- Participants That Experienced BPAR: A subset of the participants that Initiated Immunosuppression Withdrawal (ISW) and experienced biopsy-proved acute rejection (BPAR) with elevated liver function tests at the time of the biopsy were examined for this endpoint.
Arm/Group | Participants That Experienced BPAR
Number analyzed (Participants) | 35
Weeks | 13 [8.4 to 16.6]

5. Secondary Outcome: Number and Severity of Biopsies Read as Histologic Acute Rejection
Description: Number of biopsies that were diagnosed as histologic acute rejection in participants who initiated immunosuppression withdrawal by severity of rejection episode. Rejection severity (mild, moderate, severe) is based on the Banff global assessment grade according to the central pathology reading of the liver biopsy. Mild severity criteria: rejection infiltrate in a minority of triads that is generally mild and confined within the portal spaces. Moderate rejection criteria: rejection infiltrate expanding most or all of the triads. Severe rejection criteria: rejection infiltrate expanding most or all of the triads with spillover into periportal areas and moderate to severe perivenular inflammation that extends into the hepatic parenchyma and is associated with perivenular hepatocyte necrosis.
  BPAR: biopsy-proven acute rejection.
Time Frame: Time from immunosuppression withdrawal through a minimum of 36 months and maximum of 48 months of follow-up
Population: Intent-to-Treat
Measure: Number; unit: Biopsies Diagnosed as BPAR
Arm/Group | Participants That Initiated Immunosuppression Withdrawal (ISW)
Number analyzed (Participants) | 88
Biopsies Diagnosed as BPAR
  Mild | 43
  Moderate | 7
  Severe | 0

6. Secondary Outcome: Clinical Severity of Acute Rejection
Description: The clinical severity of acute rejection was descriptively analyzed using hierarchical categories, as follows:
  * Dose increase: Increase in IS dose and/or frequency but to a level less than the regimen at study entry, prior to initiating ISW
  * Reinstitution: Returning to the regimen at study entry, prior to ISW
  * Intensification: Increased IS dose compared with the dose at study entry, prior to ISW
  * Conversion: Change to different IS drug
  * Addition: Initiation of a second IS drug;
  * Corticosteroids: Administration of any intravenous or oral corticosteroids
  * Antibody (Ab) treatment: Administration of any rabbit thymoglobulin; usually with corticosteroids
Time Frame: Time from immunosuppression withdrawal through a minimum of 36 months and maximum of 48 months of follow-up
Population: Participants who experienced rejection (biopsy-proven or clinical)
Measure: Number (95% Confidence Interval); unit: Proportion
Groups:
- Participants With Adverse Events of BPAR or Clinical Rejection: All participants that initiated withdrawal were at risk for a rejection event and are included in the denominator of the proportion. Participants that had one or more adverse events of Biopsy-Proven Acute Rejection (BPAR) or Clinical Rejection and were treated with each specific treatment regimen are included in the numerator.
Arm/Group | Participants With Adverse Events of BPAR or Clinical Rejection
Number analyzed (Participants) | 88
Proportion
  Dose increase | 0.068 [0.025 to 0.143]
  Reinstitution | 0.261 [0.173 to 0.366]
  Intensification | 0.227 [0.145 to 0.329]
  Conversion | 0.011 [0 to 0.062]
  Addition | 0.023 [0 to 0.08]
  Corticosteroids | 0.364 [0.264 to 0.473]
  Ab treatment | 0 [0 to 0.041]

7. Secondary Outcome: Reason for Discontinuation of Withdrawal
Description: Reasons participants discontinued immunosuppression withdrawal, such as Biopsy Proven Acute Rejection, Chronic Rejection, Clinical Rejection, Death, Pregnancy, etc.). Only the root cause for discontinuation for each subject is presented in these results if multiple events led to discontinuation of immunosuppression withdrawal.
Time Frame: Time from start of immunosuppression withdrawal through discontinuation of withdrawal, a maximum of 52 weeks
Population: Participants who failed immunosuppression withdrawal.
Measure: Count of Participants; unit: Participants
Groups:
- Participants That Discontinued Immunosuppression Withdrawal: A subset of the Participants that Initiated Withdrawal and discontinued Immunosuppression Withdrawal (ISW) prior to completing withdrawal.
Arm/Group | Participants That Discontinued Immunosuppression Withdrawal
Number analyzed (Participants) | 33
Participants
  Biopsy Proven Acute Rejection | 30
  Clinical Rejection | 3

8. Secondary Outcome: Impact of Immunosuppression Withdrawal (ISW) on Allograft Histology
Description: The impact of ISW on allograft fibrosis using the Ishak scoring system to measure the change in fibrosis from the screening liver biopsy to the end-of-study (month-48) liver biopsy.
  In the Ishak histologic scoring system, the higher the score/stage, the more fibrosis: Scores range from 0 to 6, with 6 representing the most fibrosis: 0=No fibrosis; 1=Fibrous expansion of some portal areas, with or without short fibrous septa; 2=Fibrous expansion of most portal areas, with or without short fibrous septa; 3=Fibrous expansion of most portal areas, with occasional portal to portal bridging; 4=Fibrous expansion of portal areas with marked bridging (portal to portal) as well as portal to central; 5=Marked bridging (portal to portal and/or portal to central) with occasional nodules (incomplete cirrhosis); and 6=Cirrhosis, probable or definite.
  Decrease in score from screening (baseline) indicates improvement
Time Frame: Time from screening biopsy to end of study (month 48) biopsy
Population: Intent-to-Treat
  -Of the original 88 participants, 3 participants did not finish the study and 1 participant did not complete the final liver biopsy.
Measure: Count of Participants; unit: Participants
Groups:
- Participants That Had Both Screening and End-of-Study Biopsies: Pediatric liver transplant recipients with stable liver tests (ALT and GGT), no evidence of rejection in the preceding 2 years, and at least 4 years post-transplant, and a qualifying liver biopsy at screening underwent gradual Immunosuppression withdrawal in no less than 36 weeks and no more than 52 weeks with frequent monitoring of liver tests. All participants were followed for 48 months ensuring a minimum of 36 months of follow-up after successful Immunosuppression withdrawal.
Arm/Group | Participants That Had Both Screening and End-of-Study Biopsies
Number analyzed (Participants) | 84
Participants
  Ishak Score Change of -1 | 18
  Ishak Score Change of 0 | 43
  Ishak Score Change of 1 | 19
  Ishak Score Change of 2 | 3
  Ishak Score Change of 3 | 1

9. Secondary Outcome: Duration of Operational Tolerance
Description: Median participant duration of operational tolerance. Duration of operational tolerance is defined as the number of days that participants are not taking immunosuppression medications.
Time Frame: Time from immunosuppression withdrawal through a minimum of 36 months and a maximum of 48 months of follow-up
Population: Participants that Completed Withdrawal and were Operationally Tolerant
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Participants Deemed Tolerant by Trial Definition: Pediatric liver transplant recipients with stable liver tests (ALT and GGT), no evidence of rejection in the preceding 2 years, and at least 4 years post-transplant, and a qualifying liver biopsy at screening underwent gradual Immunosuppression withdrawal in no less than 36 weeks and no more than 52 weeks with frequent monitoring of liver tests. All participants were followed for 48 months ensuring a minimum of 36 months of follow-up after successful Immunosuppression withdrawal.
Arm/Group | Participants Deemed Tolerant by Trial Definition
Number analyzed (Participants) | 33
days | 1209.5 [1205 to 1214]

10. Secondary Outcome: Change in Immunosuppression Medication (Calcineurin Inhibitor) Dose From Start of Immunosuppression Withdrawal to the Time of Immunosuppression Withdrawal Failure
Description: The mean percent of immunosuppression (IS) dose reduction from baseline to the time of immunosuppression withdrawal failure. Immunosuppression withdrawal failure is defined as any incidence of increasing immunosuppression medications instead of completing withdrawal.
Time Frame: Time from starting immunosuppression withdrawal until immunosuppression withdrawal failure, maximum 52 weeks
Population: Intent-to-Treat who failed immunosuppression withdrawal
Measure: Mean (95% Confidence Interval); unit: percentage of dose
Groups:
- Participants That Discontinued Immunosuppression Withdrawal: A subset of the Participants that Initiated Withdrawal and discontinued Immunosuppression Withdrawal prior to completing withdrawal.
Arm/Group | Participants That Discontinued Immunosuppression Withdrawal
Number analyzed (Participants) | 33
percentage of dose | -76.1 [-80.59 to -71.63]

11. Secondary Outcome: Change in Immunosuppression Medication Dose From Study Initiation of Withdrawal to the End of the Study
Description: Change of immunosuppression (IS) dose from baseline to end of study for all participants not deemed tolerant by the trial definition either due to discontinuing IS withdrawal or completing withdrawal but not meeting the criteria for tolerance on the primary endpoint biopsy assessment.
Time Frame: Time from immunosuppression withdrawal through a minimum of 36 months and maximum of 48 months of follow-up
Population: Intent-to-Treat participants who were not operationally tolerant and who remained on the same medication throughout the study. Three subjects that were not operationally tolerant converted to alternate immunosuppression medications.
Measure: Mean (95% Confidence Interval); unit: percentage of dose
Groups:
- Participants Not Deemed Tolerant by the Trial Definition: All participants not deemed tolerant by the trial definition either due to discontinuing IS withdrawal or completing withdrawal but not meeting the criteria for tolerance on the primary endpoint biopsy.
Arm/Group | Participants Not Deemed Tolerant by the Trial Definition
Number analyzed (Participants) | 52
percentage of dose | 0.4 [-21.12 to 21.98]

12. Secondary Outcome: Change in Child Health Related Quality of Life Scores Between Tolerant and Non-tolerant Subjects
Description: Health related quality of life was measured by the PedsQL 4.0 Generic Core scale, the Multidimensional Fatigue scale, and the PedsQL 3.0 Transplant module. Change was calculated as the difference between the questionnaire completed at the initiation of withdrawal and at month 36 for the total generic score, the total fatigue score, and total transplant score. This change was calculated separately for tolerant and non-tolerant subjects. Each score ranges from 0-100, with a higher score indicating a better quality of life.
Time Frame: Time from immunosuppression withdrawal through a minimum of 36 months and maximum of 48 months of follow-up
Population: Intent-to-Treat
Measure: Mean (95% Confidence Interval); unit: Quality of Life Scores on a Scale
Groups:
- Participants Were Operationally Tolerant: Participants that Completed Withdrawal and were Operationally Tolerant
- Participants Who Were Not Operationally Tolerant: Participants who were not operationally tolerant.
Arm/Group | Participants Were Operationally Tolerant | Participants Who Were Not Operationally Tolerant
Number analyzed (Participants) | 33 | 55
Quality of Life Scores on a Scale
  Total Generic Score | 3.4 [-0.8 to 7.7] | 1.2 [-2.1 to 4.5]
  Total Fatigue Score | 5.0 [1.2 to 8.8] | 2.0 [-3.9 to 7.8]
  Total Transplant Score | 5.7 [1.7 to 9.8] | 0.9 [-2.5 to 4.2]

ADVERSE EVENTS:
Time Frame: Time of enrollment through end of study participation (e.g., up to 48 months).
Description: Safety tables include N=161 participants,inclusive of those that were not eligible (N=73) and eligible (N=88) to proceed with immunosuppression withdrawal (ISW):
  * Adverse events (AEs) were collected from the time of enrollment (i.e., assessment for eligibility to initiate immunosuppression withdrawal [ISW]) through the end of study participation;
  * Prior to initiating ISW, only AEs temporally related to study procedures were collected; and,
  * All AEs were collected ≥initiation of ISW.
Groups:
- All Enrolled Participants: Pediatric liver transplant recipients with stable liver function tests, no evidence of rejection in the past 2 years, and at least 4 years post-transplant, and a qualifying liver biopsy at screening underwent gradual Immunosuppression withdrawal in no less than 36 weeks and no more than 52 weeks with frequent monitoring of liver tests. All participants were followed for 48 months ensuring a minimum of 36 months of follow-up after successful Immunosuppression withdrawal.
Arm/Group | All Enrolled Participants
All-Cause Mortality (participants affected / at risk) | 0/161
Serious Adverse Events (participants affected / at risk) | 23/161
Other Adverse Events (participants affected / at risk) | 87/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Participants (N=161)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 2 (2)
Transplant rejection (Immune system disorders) | 3 (4)
Cellulitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 2 (5)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 1 (1)
Varicella (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 2 (2)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Oppositional defiant disorder (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Participants (N=161)
Abdominal pain (Gastrointestinal disorders) | 17 (25)
Diarrhoea (Gastrointestinal disorders) | 16 (21)
Vomiting (Gastrointestinal disorders) | 9 (12)
Influenza like illness (General disorders) | 16 (36)
Pyrexia (General disorders) | 14 (19)
Hypersensitivity (Immune system disorders) | 10 (11)
Transplant rejection (Immune system disorders) | 37 (43)
Ear infection (Infections and infestations) | 13 (26)
Gastroenteritis (Infections and infestations) | 14 (17)
Gastroenteritis viral (Infections and infestations) | 21 (28)
Influenza (Infections and infestations) | 14 (16)
Nasopharyngitis (Infections and infestations) | 35 (140)
Pharyngitis streptococcal (Infections and infestations) | 16 (20)
Sinusitis (Infections and infestations) | 12 (24)
Upper respiratory tract infection (Infections and infestations) | 21 (36)
Viral infection (Infections and infestations) | 19 (39)
Liver function test abnormal (Investigations) | 24 (39)
Headache (Nervous system disorders) | 17 (37)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (21)
Rash (Skin and subcutaneous tissue disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No